CLINICAL TRIAL: NCT05263466
Title: Dosimetry and Immunohistochemistry Study to Establish Radiolabelled PSMA as a Potential Target in Glioma Treatment
Brief Title: Establishing Radiolabelled PSMA as a Target for Glioma Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 306945
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain tumour patients (Experimental): Patients will be those undergoing routine care of primary brain tumours. Study group patients will undergo additional PET-MRI examination and biopsies in addition to the standard of care.
  Interventions: Diagnostic Test: PET-MRI; Procedure: Brain tumour biopsy

INTERVENTIONS:
Diagnostic Test: PET-MRI — For the diagnostic imaging aspect included in this pilot study, [68Ga]PSMA-11 will be used. This is a peptidomimetic agent with a covalently bound chelator (HBED-CC) that is FDA-approved in prostate cancer imaging. We will use PET-MRI to visualise a) the concentration and b) the distribution of this tracer to establish a functional map of primary brain tumour activity
Procedure: Brain tumour biopsy — All patients included in our study will undergo stereotactic surgery for biopsy/resection of the tumour as part of the standard of care at KCH. During this study we will not vary from the surgical standard of care for primary brain tumours and will only extend the surgery time due to additional stereotactic biopsies (an additional 3 biopsies increasing the time of the operation by ~30 minutes). Professor Ashkan (KCH) has defined the additional surgical risk of performing these biopsies to be ~0%, since targeted biopsies will only be taken within the tumour just before resection. The stereotactic biopsy may be targeted to areas of high [68Ga]PSMA SUV within the tumour as defined by the PET MRI scan.

SUMMARY:
A study is being performed to observe whether a novel type of brain imaging using a technique called PET-MRI may provide useful information in the 'mapping' of adult primary brain tumours. It employs a radiolabelled molecule targeting a particular molecule called PSMA which is hypothesised to be a marker of aggression in primary brain tumours. 'Mapping' of the concentration and distribution of this molecule within brain tumours via PET-MRI may provide vital clinical information regarding the extent and timing of treatment.

DETAILED DESCRIPTION:
One potential avenue of high grade glioma treatment involves a 'theranostic' radiotherapeutic approach. This consists of two stages: firstly, a particular protein expressed specifically by the tumour is radiolabelled with a targeted radioligand emitting gamma radiation, enabling confirmation of the presence, concentration and distribution of this target protein (diagnostic stage). Following this, a similar ligand is this time attached to an alpha or beta-emitter, enabling targeted tumour destruction (therapeutic stage).

There is growing, but limited, evidence that prostate specific membrane antigen (PSMA) is strongly and specifically expressed in high grade glioma and may be a potential theranostic target [Wernicke 2011, Unterrainer 2017]. It has already been used extensively as a theranostic target in metastatic prostate cancer, demonstrating safety and efficacy in this condition [Abou et al 2020].

The clinical outcomes shown in prostate cancer, along with evidence of PSMA expression in high grade glioma, led the study team to convene an Incubator Day with a group of experts to explore the possibility of developing a PSMA-targeting theranostic agent in high grade glioma. Expertise included PSMA theranostics (Prof Lewington), neuro-oncology (Dr Brazil, Guy's and St Thomas' Hospital (GSTT)), neurosurgery (Prof Ashkan, King's College Hospital (KCH)), neuropathology (Prof Al-Sarraj, KCH), neuroradiology (Dr Booth, KCH) PSMA PET imaging (Prof Gary Cook and Prof Alexander Hammers GSTT/KCL), nuclear physics (Prof Paul Marsden GSTT/KCL), and PSMA radiopharmaceutical chemistry (Prof Blowers, KCL).

It was concluded that a PSMA-targeting theranostic agent has the potential to be a safe and effective treatment for high grade glioma. The regulatory pathway should be eased enormously by the precedent of use in prostate cancer, which would obviate the need for pre-clinical studies.

This approach was conditional upon two objectives:

1. Perform a series of five [68Ga]PSMA PET scans for dosimetry analysis and assessment of the retention of the tracer in the tumour (Using GSTT/KCL PET/MRI) prior to biopsy, at the same time as the patient's routine brain tumour imaging series. At time of recurrence a further [68 Ga]PSMA PET-MRI scan may be performed in each patient (depending on whether or not recurrence occurs during the study period) to assess for change in the standardised uptake value (SUV).
2. Performing immunohistochemical analysis on high grade glioma specimens (prospectively in patients enrolled in this study with additional retrospective samples), in order to replicate published evidence on the expression of PSMA in such tumours, and also to demonstrate in the prospective cohort, a correlation between imaging detection of [68 Ga]PSMA and histopathological detection in stereotactic brain tumour biopsy samples (Using KCH neuropathology facilities).

ELIGIBILITY:
Inclusion Criteria:

* Individuals of 18 years or older
* Referred for surgery (resection or biopsy) of presumed high grade primary brain tumour (based on imaging features of aggression e.g. perfusion imaging, diffusion restriction etc.). As standard, all patients will have had a full body CT and other investigations to rule out metastatic disease (this has a very high negative predictive value).
* Written informed consent

Exclusion Criteria:

* Patient already enrolled in a drug trial
* Contra-indication for MRI contrast
* Contra-indication for radiotracer
* Inability to give consent
* Patient is pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of the PET-MRI PSMA signal intensity (arbitrary units) and glioma protein concentration (g/L) in a 1 x 1 x 1 cm region of interest (R value) | 5 years
  PET-MRI signal will be recorded from different regions of interest within a glioma where stereotactic surgical biopsies taken and protein concentration determined.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Booth, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louis DN, Wesseling P, Aldape K, Brat DJ, Capper D, Cree IA, Eberhart C, Figarella-Branger D, Fouladi M, Fuller GN, Giannini C, Haberler C, Hawkins C, Komori T, Kros JM, Ng HK, Orr BA, Park SH, Paulus W, Perry A, Pietsch T, Reifenberger G, Rosenblum M, Rous B, Sahm F, Sarkar C, Solomon DA, Tabori U, van den Bent MJ, von Deimling A, Weller M, White VA, Ellison DW. cIMPACT-NOW update 6: new entity and diagnostic principle recommendations of the cIMPACT-Utrecht meeting on future CNS tumor classification and grading. Brain Pathol. 2020 Jul;30(4):844-856. doi: 10.1111/bpa.12832. Epub 2020 Apr 19. PMID 32307792
- [Background] Wernicke AG, Edgar MA, Lavi E, Liu H, Salerno P, Bander NH, Gutin PH. Prostate-specific membrane antigen as a potential novel vascular target for treatment of glioblastoma multiforme. Arch Pathol Lab Med. 2011 Nov;135(11):1486-9. doi: 10.5858/arpa.2010-0740-OA. PMID 22032578
- [Background] Unterrainer M, Niyazi M, Ruf V, Bartenstein P, Albert NL. The endothelial prostate-specific membrane antigen is highly expressed in gliosarcoma and visualized by [68Ga]-PSMA-11 PET: a theranostic outlook for brain tumor patients? Neuro Oncol. 2017 Nov 29;19(12):1698-1699. doi: 10.1093/neuonc/nox172. No abstract available. PMID 29045711
- [Background] Abou D, Benabdallah N, Jiang W, Peng L, Zhang H, Villmer A, Longtine MS, Thorek DLJ. Prostate Cancer Theranostics - An Overview. Front Oncol. 2020 Jun 5;10:884. doi: 10.3389/fonc.2020.00884. eCollection 2020. PMID 32582550